CLINICAL TRIAL: NCT02291952
Title: Development of Countermeasures Against Adverse Metabolic Effects of Shift Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Frank AJL Scheer, PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01HL118601 (NIH)
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Circadian Dysregulation
Keywords: Circadian Misalignment, Forced Desynchrony, Metabolism, Meal-timing, Circadian
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): During Forced Desynchrony sleep and wake will occur at different circadian phases, while meals are restricted to the biological day.
  Interventions: Behavioral: Meal schedule
- Control (Other): During Forced Desynchrony sleep and wake, as well as meals, will occur at different circadian phases.
  Interventions: Behavioral: Meal schedule

INTERVENTIONS:
Behavioral: Meal schedule

SUMMARY:
The goal of this application is to determine whether changing the timing of food intake prevents the adverse metabolic effects of circadian misalignment.

DETAILED DESCRIPTION:
Shift work is associated with circadian misalignment and an increased risk for the development diabetes, obesity, and cardiovascular disease. This research will determine whether changing the feeding schedule can prevent metabolic alterations that can lead to the abovementioned disorders. This research will provide mechanistic insight and may provide a novel therapeutic approach against the increased risk for diabetes, obesity, and cardiovascular disease among shift workers.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 29.9 kgm-2
* Healthy adults with regular sleep-wake timing
* Non-smokers
* Completion of medical and psychological screening tests
* Able to spend 14 consecutive days in the sleep laboratory

Exclusion Criteria:

* BMI <18.5 or > 29.9 kgm-2
* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Donating blood within past 8 weeks
* Worked night or rotating shift work within past 3 years
* Hearing impairment
* Drug or alcohol dependency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Change in plasma leptin levels across sleep/wake cycle | During circadian alignment (Day 7) and circadian misalignment (Day 10-11)
  Frequent blood samples
Change in circadian profile of plasma leptin | During constant routine before forced desynchrony (Days 3-4) and constant routine after forced desynchrony (Days 12-13)
  Frequent blood samples
Change in glucose tolerance | During circadian alignment (Day 7) and circadian misalignment (Day 10-11)
  Frequent blood samples before and after standardized meals
Change in circadian profile of plasma glucose levels | During circadian alignment (Day 7) and circadian misalignment (Day 10-11)
  Frequent blood samples
Change in plasma insulin levels after standardized test meal | During circadian alignment (Day 7) and circadian misalignment (Day 10-11)
  Frequent blood samples before and after standardized meals
Change in circadian profile of plasma insulin levels | During circadian alignment (Day 7) and circadian misalignment (Day 10-11)
  Frequent blood samples

SECONDARY OUTCOMES:
o Change in circadian phase markers, such as from core body temperature, melatonin, and cortisol | Core temperature and frequent blood samples
  Core temperature sensor throughout protocol, days 1-14. Frequent blood samples during constant routine before forced desynchrony (Days 3-4) and constant routine after forced desynchrony (Days 12-13)
Changes circadian rhythm in resting energy expenditure | During constant routine before forced desynchrony (Days 3-4) and constant routine after forced desynchrony (Days 12-13)
  Indirect calorimetry
Change in hunger and appetite, mood, and cognitive performance | Tests taken throughout the protocol, days 1-14
  Subjective hunger ratings and cognitive tests performed via computer interface
Changes in microbiota, gene expression, epigenetic or proteomic markers | samples taken during forced desychrony (days 7-11) and the constant routine protocols (days 3-4 and 11-13)
  Frequent blood samples and saliva samples
Changes in sleep | sleep periods following day 1, days 6-7 and days 10-11
  Polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chellappa SL, Engen PA, Naqib A, Qian J, Vujovic N, Rahman N, Green SJ, Garaulet M, Keshavarzian A, Scheer FAJL. Proof-of-principle demonstration of endogenous circadian system and circadian misalignment effects on human oral microbiota. FASEB J. 2022 Jan;36(1):e22043. doi: 10.1096/fj.202101153R. PMID 34861073